CLINICAL TRIAL: NCT00947050
Title: Prompt Human Coronary Collateral Vasomotor Function Induced by Dynamic Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: University hospital Bern, Cardiology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14/05
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Artery Disease
Keywords: CAD; prompt physical exercise; collateral function
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rest first (Active Comparator): rest first, cfi, exercise, cfi
  Interventions: Other: dynamic physical exercise
- exercise first (Active Comparator): ex first
  Interventions: Other: dynamic physical exercise

INTERVENTIONS:
Other: dynamic physical exercise — dynamic supine bicycle exercise for 6 minutes
  Other Names: rest first; ex first

SUMMARY:
The purpose of this study in humans with stable coronary artery disease (CAD) treatable by PCI (percutaneous coronary intervention) is to evaluate if dynamic physical exercise leads to an instantaneous improvement of coronary collateral function.

DETAILED DESCRIPTION:
The existence of coronary collateral vessels and their benefit against cardiac events have been recognized for many years, but their functional capacity in response to physical exercise has partially remained elusive. Via endothelial shear stress, the fundamental stimulus for collateral development, exercise theoretically leads to collateral vasodilation and recruitment by an increase in heart rate and blood pressure during exercise. Moreover, the phenomenon of "walking through angina" indicates that collateral function and physical activity are related and their interaction is of clinical relevance.

The purpose of the present study in humans with stable coronary artery disease was to assess the instantaneous response of coronary collateral function to dynamic physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or 18 years old
* 1- to 3-vessel coronary artery disease (CAD)
* Stable angina pectoris
* At least 1 stenotic lesion suitable for PCI
* Negative Allen-test
* Written informed consent to participate in the study

Exclusion Criteria:

* Patients admitted as emergencies
* Acute myocardial infarction
* Unstable CAD
* Q-wave myocardial infarction in the area undergoing CFI measurement
* CAD treated best by CABG
* Severe valve disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change of collateral flow index (CFI, no unit) during exercise (E) compared to CFI at rest (R). | 6 minutes

SECONDARY OUTCOMES:
Correlation of collateral flow index change and maximal workload. | 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Gloekler, MD, Principal Investigator — University of Bern; Mario Togni, MD, Principal Investigator — University of Bern; Pascal Meier, MD, Principal Investigator — University of Bern; Christian Seiler, MD,Prof., Study Chair — University of Bern; Stefano de Marchi, MD, Principal Investigator — Univerity of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Togni M, Gloekler S, Meier P, de Marchi SF, Rutz T, Steck H, Traupe T, Seiler C. Instantaneous coronary collateral function during supine bicycle exercise. Eur Heart J. 2010 Sep;31(17):2148-55. doi: 10.1093/eurheartj/ehq202. Epub 2010 Jun 28. PMID 20584776